CLINICAL TRIAL: NCT03045679
Title: The Evidence of One-anastomosis Gastric Bypass/Mini-Gastric Bypass Versus Roux-en Y Gastric Bypass in Metabolic Surgery - a Prospective Randomized Controlled Trial
Brief Title: One-anastomosis Gastric Bypass/Mini-Gastric Bypass Versus Roux-en Y Gastric Bypass
Acronym: MGBvsRYGB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Hospital changed in 2019, no recruitment performed
Sponsor: Sana Klinikum Offenbach (Other)
Responsible Party: Principal Investigator, Sonja Chiappetta, MD, Principal investigator: Dr. Sonja Chiappetta, Sana Klinikum Offenbach
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FF 74/2016
Record Dates: First submitted 2017-02-05; First posted 2017-02-07 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Obesity
Keywords: Roux-en Y gastric bypass; One-anastomosis gastric bypass; Mini-gastric bypass; metabolic surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled trial: RYGB (group A) vs OAGB/MGB (group B)
Who Masked: Investigator
Masking Description: envelope randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RYGB-group (Experimental): Patients who undergo laparoscopic RYGB (150 cm alimentary limb, 50 cm biliopancreatic limb) as a primary surgery in obesity surgery; n = 50
  Interventions: Other: RYGB
- OAGB/MGB-group (Experimental): Patients who undergo laparoscopic OAGB/MGB (200 cm biliopancreatic limb) as a primary surgery in obesity surgery; n = 50
  Interventions: Other: OAGB/MGB

INTERVENTIONS:
Other: RYGB — laparoscopic RYGB
  Arms: RYGB-group
Other: OAGB/MGB — laparoscopic OAGB/MGB
  Arms: OAGB/MGB-group

SUMMARY:
The aim of this prospective randomized controlled trial is to compare the two procedures One-anastomosis gastric Bypass/Mini-gastric Bypass (OAGB/MGB) and Roux-en Y gastric bypass (RYGB) in relation to intraoperative and postoperative complications (classification of Clavien-Dindo), mortality, metabolic impact (remission of type 2 diabetes mellitus, hypertonus, gastro-esophageal reflux disease, sleep apnea, dyslipidemia, quality of life, operation time, postoperative excess weight loss, malnutrition and re-do/revisonal surgery.

DETAILED DESCRIPTION:
OAGB/MGB is gaining popularity as a primary surgical treatment for morbid obesity due to reduced operation time, a shorter learning curve, better weight loss, higher metabolic impact and fewer major complications compared to RYGB.

In this prospective randomized controlled trial we want to compare OAGB/MGB and RYGB with a FU of up to 24 month.

Patients with indication for gastric bypass get randomized in group A (RYGB, n = 50) or B (OAGB/MGB, n = 50). FU is performed 1, 3, 6, 12 and 24 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. primary obesity surgery and indication for gastric bypass
2. age: 18 - 65 years
3. BMI > 40 kg/m² or BMI > 35 kg/m² with obesity related comorbidities
4. informed consent

Exclusion Criteria:

1. obesity surgery in the anamnesis
2. visceral surgery in the anamnesis (excluding appendectomy and cholecystectomy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
complications | up to 2 years after surgery
  complications classified next to Clavien-Dindo

SECONDARY OUTCOMES:
mortality | up to 2 years after surgery
  death up to 2 years after surgery
remission of type 2 diabetes mellitus | up to 2 years after surgery
  HbA1c < 6.5% without medication
remission of hypertonus | up to 2 years after surgery
  blood pressure < 140/90 mmHg without medication
gastro-esophageal reflux disease | up to 2 years after surgery
  GERD-HRGL Heartburn Scale
remission of sleep apnea | up to 2 years after surgery
  presence/absence of CPAP
remission of hypertrigliceridemia | up to 2 years after surgery
  triglyceride < 200mg/dl without medication
remission of hypercholesterinemia | up to 2 years after surgery
  cholesterin < 155 mg/dl without medication
quality of life questionnaire | up to 2 years after surgery
  changing in quality of life measured by questionnaire
weight loss | up to 2 years after surgery
  postoperative excess weight loss in %
operation time | operation time during surgery in minutes
  operation time during surgery in minutes
malnutrition 1 | up to 2 years after surgery
  postoperative malnutrition: protein < 64 g/l
malnutrition 2 | up to 2 years after surgery
  postoperative malnutrition: albumin < 35 g/l
malnutrition 3 | up to 2 years after surgery
  postoperative malnutrition: ferritin (< 30 µg/l)
malnutrition 4 | up to 2 years after surgery
  postoperative malnutrition: vitamin E < 12 µmol/l
malnutrition 5 | up to 2 years after surgery
  postoperative malnutrition: vitamin K < 90 ng/l
malnutrition 6 | up to 2 years after surgery
  postoperative malnutrition: vitamin 25-OH- Vitamin D3 < 50 nmol/l
malnutrition 7 | up to 2 years after surgery
  postoperative malnutrition: vitamin A < 1.05 µmol/l
malnutrition 8 | up to 2 years after surgery
  postoperative malnutrition: vitamin B12 < 145 pmol/l
revisional surgery | up to 2 years after surgery
  revisional surgery during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Chiappetta, MD, Study Chair — Sana Klinikum Offenbach
Locations (1):
- Sana Klinikum Offenbach, Offenbach, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chevallier JM, Arman GA, Guenzi M, Rau C, Bruzzi M, Beaupel N, Zinzindohoue F, Berger A. One thousand single anastomosis (omega loop) gastric bypasses to treat morbid obesity in a 7-year period: outcomes show few complications and good efficacy. Obes Surg. 2015 Jun;25(6):951-8. doi: 10.1007/s11695-014-1552-z. PMID 25585612
- [Result] Jammu GS, Sharma R. A 7-Year Clinical Audit of 1107 Cases Comparing Sleeve Gastrectomy, Roux-En-Y Gastric Bypass, and Mini-Gastric Bypass, to Determine an Effective and Safe Bariatric and Metabolic Procedure. Obes Surg. 2016 May;26(5):926-32. doi: 10.1007/s11695-015-1869-2. PMID 26337694
- [Result] Musella M, Apers J, Rheinwalt K, Ribeiro R, Manno E, Greco F, Cierny M, Milone M, Di Stefano C, Guler S, Van Lessen IM, Guerra A, Maglio MN, Bonfanti R, Novotna R, Coretti G, Piazza L. Efficacy of Bariatric Surgery in Type 2 Diabetes Mellitus Remission: the Role of Mini Gastric Bypass/One Anastomosis Gastric Bypass and Sleeve Gastrectomy at 1 Year of Follow-up. A European survey. Obes Surg. 2016 May;26(5):933-40. doi: 10.1007/s11695-015-1865-6. PMID 26341086
- [Result] Guenzi M, Arman G, Rau C, Cordun C, Moszkowicz D, Voron T, Chevallier JM. Remission of type 2 diabetes after omega loop gastric bypass for morbid obesity. Surg Endosc. 2015 Sep;29(9):2669-74. doi: 10.1007/s00464-014-3987-7. Epub 2015 Jan 1. PMID 25552228
- [Result] Lee WJ, Yu PJ, Wang W, Chen TC, Wei PL, Huang MT. Laparoscopic Roux-en-Y versus mini-gastric bypass for the treatment of morbid obesity: a prospective randomized controlled clinical trial. Ann Surg. 2005 Jul;242(1):20-8. doi: 10.1097/01.sla.0000167762.46568.98. PMID 15973097